CLINICAL TRIAL: NCT03018522
Title: S100B Protein as Predictor of Cognitive Dysfunction After Robot-assisted Radical Prostatectomy: A Prospective Observational Study
Brief Title: S100B Protein and Postoperative Cognitive Dysfunction
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: AntalyaTRH14
Record Dates: First submitted 2017-01-09; First posted 2017-01-12 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Postoperative cognitive dysfunction — Neuropsychological tests of all patients will conduct on the one day prior to surgery, the 7th day after surgery, and the 3rd month after surgery

SUMMARY:
Primary aim of this study is to evaluate the association between postoperative cognitive dysfunction and increased serum levels of S100B protein after robot-assisted laparoscopic radical prostatectomy.

DETAILED DESCRIPTION:
The neurocognitive assessment protocol will design to evaluate general cognitive function and identify patients with cognitive dysfunction. Neuropsychological tests of all patients will conduct on the one day prior to surgery, the seventh day after surgery, and the 3rd month after surgery, respectively. According to a consensus statement, cognitive function will assess using a battery of seven neuropsychological tests: Rey Auditory Verbal Learning Test (delayed recall), Trail Making Test (Parts A and B), Digit Span Test (forward and backward), and Grooved Pegboard Test (dominant and non-dominant hands). To determine a normal reference value of cognitive functions, a group of 20 healthy individuals appropriately selected with respect to sex, age and education level without any significant mental or somatic disorders and without operation were recruited as a control group. To determine the cognitive dysfunction, baseline score or time measurement were subtracted from test score and the difference was divided by the standard deviation of the score in the control group. The result was called the Z score. Z score was calculated for each test and, POCD was defined as a Z score greater than 1.96 in at least two of the seven tests, and/or a combined Z score greater than 1.96.

Serum levels of S100B protein will obtain from venous blood samples collected before surgery, after anesthesia induction, at 30 min and 24 h after surgery.

ELIGIBILITY:
Inclusion Criteria:

* over 50 years old
* scheduled for robotic-assisted laparoscopic radical prostatectomy
* the body mass index ranged from 18 kg/m2 to 25 kg/m2
* American Society of Anesthesiologists class I, II or III

Exclusion Criteria:

* Patients with previous neurological deficit (symptomatic stroke, hemorrhage, transient ischemic attack)
* other neurologic disorders (epilepsy, trauma, intra- or extracranial malignancy)
* psychiatric diseases (schizophrenia, or depressive disorder)
* alcoholism or any other drug dependence
* serious hearing or visual impairment

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults between 50 and 90 years of age with robot assisted laparoscopic radical prostatectomy , were selected in the study.
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-11-24 (Actual); Study Completion 2018-02-14 (Actual)

PRIMARY OUTCOMES:
Score in Neuropsychological Tests | Change from neuropsychological test scores at 3 months.
  This assessment will be applied before surgery, and 7 days and 3 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Nilgun Kavrut Ozturk, M.D., Study Director — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Department of Anesthesiology and Reanimation, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva FP, Schmidt AP, Valentin LS, Pinto KO, Zeferino SP, Oses JP, Wiener CD, Otsuki DA, Tort AB, Portela LV, Souza DO, Auler JO Jr, Carmona MJ. S100B protein and neuron-specific enolase as predictors of cognitive dysfunction after coronary artery bypass graft surgery: A prospective observational study. Eur J Anaesthesiol. 2016 Sep;33(9):681-9. doi: 10.1097/EJA.0000000000000450. PMID 27433840
- [Background] Tomaszewski D. Biomarkers of Brain Damage and Postoperative Cognitive Disorders in Orthopedic Patients: An Update. Biomed Res Int. 2015;2015:402959. doi: 10.1155/2015/402959. Epub 2015 Aug 31. PMID 26417595
- [Background] Chen K, Wei P, Zheng Q, Zhou J, Li J. Neuroprotective effects of intravenous lidocaine on early postoperative cognitive dysfunction in elderly patients following spine surgery. Med Sci Monit. 2015 May 15;21:1402-7. doi: 10.12659/MSM.894384. PMID 25975969
- [Background] van Munster BC, Korevaar JC, Korse CM, Bonfrer JM, Zwinderman AH, de Rooij SE. Serum S100B in elderly patients with and without delirium. Int J Geriatr Psychiatry. 2010 Mar;25(3):234-9. doi: 10.1002/gps.2326. PMID 19575407
- [Derived] Kavrut Ozturk N, Kavakli AS, Arslan U, Aykal G, Savas M. [S100B level and cognitive dysfunction after robotic-assisted laparoscopic radical prostatectomy procedures: a prospective observational study]. Braz J Anesthesiol. 2020 Nov-Dec;70(6):573-582. doi: 10.1016/j.bjan.2020.06.006. Epub 2020 Oct 15. PMID 33213866